CLINICAL TRIAL: NCT04121767
Title: Safety and Efficacy of Edoxaban Versus Warfarin in Patients Undergoing a Thoracoscopic Ablation for Persistent Atrial Fibrillation
Brief Title: Safety and Efficacy of Edoxaban in Thoracoscopic Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Dong Seop Jeong, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: samsungmc_TTA_edoxaban
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation; Anticoagulants and Bleeding Disorders
Keywords: atrial fibrillation; thoracoscopic ablation; anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Hemostatic Disorders | interventions — edoxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban group (Experimental): patients prescribed edoxaban after thoracoscopic ablation during window period to prevent stroke
  Interventions: Drug: Edoxaban
- Warfarin group (Active Comparator): patients prescribed warfarin after thoracoscopic ablation during window period to prevent stroke
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Edoxaban — oral edoxaban 60mg once daily for 3 months
  Other Names: Savaysa
  Arms: Edoxaban group
Drug: Warfarin — oral warfarin once daily for 3 months according to prothrombin time
  Other Names: Coumadin
  Arms: Warfarin group

SUMMARY:
The aim of this study is to compare the safety and efficacy of edoxaban and warfarin for prevention of stroke during a 6-month follow up after total thoracoscopic ablation.

DETAILED DESCRIPTION:
In Korea, 5% of patients older than 65 years and 10% of patients older than 80 have a history of atrial fibrillation (AF), which is often associated with sudden death and stroke. Medication and percutaneous radiofrequency catheter ablation are commonly used treatment modalities. Pharmacotherapy is primarily symptomatic treatment; moreover, the effect of conversion to a normal rhythm is minimal, and mainly aimed at stabilizing heart rate. Catheter ablation is associated with a high incidence of recurrence in chronic AF, and it is difficult to treat left atrial appendage, thereby preventing discontinuation of anticoagulation therapy post procedure. Thoracoscopic ablation is known to be a less invasive and more effective modality to treat patients with chronic atrial fibrillation. However, anticoagulation therapy is mandatory in the early postoperative period due to intracardiac thromboembolism associated with atrial stunning despite conversion to a sinus rhythm and resection of the left atrial appendage. Further investigation would be required to assess the efficacy and safety of novel oral anticoagulants such as edoxaban compared to that of warfarin for stroke prevention during the early postoperative period (6 months) after a thoracoscopic procedure. The need to maintain a constant level of blood coagulation and the potential development of complications such as hemorrhages are drawbacks associated with the use of warfarin. While novel oral anticoagulants such as edoxaban do have a role in atrial fibrillation, data regarding their effectiveness and incidence of complications after arrhythmia surgery do not exist. In this study, we will compare warfarin and edoxaban with respect to safety and efficacy, after they are used for 6 months following thoracoscopic ablation in patients with chronic atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older (not exceed 80 years old).
2. Elective thoracoscopic ablation.
3. Presence of atrial fibrillation (paroxysmal, persistent, long-standing persistent).

Exclusion Criteria:

1. Chronic obstructive pulmonary disease (COPD).
2. History of pulmonary tuberculosis.
3. Other cardiac comorbidities including valvular disease, coronary artery disease.
4. Congenital heart anomalies except for atrial septal defect.
5. Known, clinically important anemia or thrombocytopenia.
6. Pregnancy or lactation.
7. Malignancy.
8. Intracardiac mass or thrombus
9. Life expectancy less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Postoperative stroke | 6 months
  Number of patients showing thromboembolic neurologic complication after thoracoscopic ablation

SECONDARY OUTCOMES:
Postoperative bleeding | 6 months
  Number of patients showing bleeding events due to anticoagulation after thoracoscopic ablation
Postoperative pericarditis | 6 months
  Number of patients showing pericarditis requiring readmission after thoracoscopic ablation

CONTACTS AND LOCATIONS:
Overall Officials: Dong Seop Jeong, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea